CLINICAL TRIAL: NCT03352297
Title: Rejuvenation of Post Burn Scars on the Face With Unfiltered Nanofat Injection
Brief Title: Nanofat in Post Burn Scars on the Face
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Muhammad Mustehsan Bashir, Associate Professor, King Edward Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 249/PLS/MHL
Record Dates: First submitted 2017-11-15; First posted 2017-11-24 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Burn Scar
Keywords: Post burn scar face; Unfiltered nanofat; Adipose tissue growth factors; Adipose stem cells; POSAS; Image J; Face
MeSH Terms: conditions — Facies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Unfiltered Nanofat Graft — Nanofat created from microfat, skipping the filtration step. Intradermal and subdermal injections in post burn scars on the face.

SUMMARY:
Quasi-Experimental Study: Unfiltered Nanofat Injected into Postburn Facial Scars Number of Patients: 48 Outcome Assessed on POSAS And with Imaje J Scanning Preop And Postop Statistical Comparison of Scar Done

DETAILED DESCRIPTION:
Objective: To compare the quality of post burn facial scars before and after injection of unfiltered nanofat.

Place and Duration of Study: Plastic Surgery Department, Mayo Hospital, Lahore, from January 2016 to December 2016.

Methodology: 48 patients with post burn facial scars were included, age range 4 to 32 years with Fitzpatrick skin types between 3 and 4. Patients with hypertrophic scars, contractures or keloids were excluded. Scars were assessed by a senior plastic surgeon and the patient on the POSAS. Fat was harvested from the abdomen and/or thighs with a 3 mm multi-port liposuction cannula (containing several sharp side holes of 1 mm) using Coleman's technique, emulsified, and transferred into 1 ml Leur lock syringes for injection into the subdermal or intradermal plane. Final follow up was scheduled at 6 months and scar was rated by the patient and the same surgeon on the POSAS. Pre and post op scar scores were compared and p-values calculated.

ELIGIBILITY:
Inclusion Criteria:

* Post burn scars on the face
* Fitzpatrick skin types between 3 and 4

Exclusion Criteria:

* Hypertrophic scars
* Contractures
* Keloids

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Rejuvenation of post burn scars on the face with unfiltered nanofat injection | 1 year
  Pre and post-operative POSAS score

CONTACTS AND LOCATIONS:
Overall Officials: Saadia Jan, FRCS ed, FCPS, Principal Investigator — King Edward Medical University Lahore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neuber G. Über die Wiederanheilung vollständig vom Körper getrennter, die ganze Fettschicht enthaltender Hautstücke. Zentralblatt Chir. 1893;30:16
- [Background] Illouz YG. Body contouring by lipolysis: a 5-year experience with over 3000 cases. Plast Reconstr Surg. 1983 Nov;72(5):591-7. doi: 10.1097/00006534-198311000-00001. PMID 6622564
- [Background] Stuschke M, Budach V, Sack H. Radioresponsiveness of human glioma, sarcoma, and breast cancer spheroids depends on tumor differentiation. Int J Radiat Oncol Biol Phys. 1993 Oct 20;27(3):627-36. doi: 10.1016/0360-3016(93)90389-d. PMID 8226158
- [Background] Coleman SR. Structural fat grafts: the ideal filler? Clin Plast Surg. 2001 Jan;28(1):111-9. PMID 11248861
- [Background] Zuk PA, Zhu M, Mizuno H, Huang J, Futrell JW, Katz AJ, Benhaim P, Lorenz HP, Hedrick MH. Multilineage cells from human adipose tissue: implications for cell-based therapies. Tissue Eng. 2001 Apr;7(2):211-28. doi: 10.1089/107632701300062859. PMID 11304456
- [Result] Tonnard P, Verpaele A, Peeters G, Hamdi M, Cornelissen M, Declercq H. Nanofat grafting: basic research and clinical applications. Plast Reconstr Surg. 2013 Oct;132(4):1017-1026. doi: 10.1097/PRS.0b013e31829fe1b0. PMID 23783059
- [Result] Lo Furno D, Tamburino S, Mannino G, Gili E, Lombardo G, Tarico MS, Vancheri C, Giuffrida R, Perrotta RE. Nanofat 2.0: experimental evidence for a fat grafting rich in mesenchymal stem cells. Physiol Res. 2017 Sep 22;66(4):663-671. doi: 10.33549/physiolres.933451. Epub 2017 Apr 12. PMID 28406706
- [Result] Goisis M, Stella E, Di Petrillo A, Rosset L. Nanofat Grafting Compared to Hyaluronic Acid and PRP Treatment of the Lower Lid and Tear Trough: Clinical Outcome. JSM Ophthalmology. 2015;3:1027
- [Result] Jaspers MEH, Brouwer KM, van Trier AJM, Groot ML, Middelkoop E, van Zuijlen PPM. Effectiveness of Autologous Fat Grafting in Adherent Scars: Results Obtained by a Comprehensive Scar Evaluation Protocol. Plast Reconstr Surg. 2017 Jan;139(1):212-219. doi: 10.1097/PRS.0000000000002891. PMID 27632398
- [Result] Mailey B, Saba S, Baker J, Tokin C, Hickey S, Wong R, Wallace AM, Cohen SR. A comparison of cell-enriched fat transfer to conventional fat grafting after aesthetic procedures using a patient satisfaction survey. Ann Plast Surg. 2013 Apr;70(4):410-5. doi: 10.1097/SAP.0b013e31827e5353. PMID 23486128
- [Result] Kim JH, Jung M, Kim HS, Kim YM, Choi EH. Adipose-derived stem cells as a new therapeutic modality for ageing skin. Exp Dermatol. 2011 May;20(5):383-7. doi: 10.1111/j.1600-0625.2010.01221.x. Epub 2011 Feb 28. PMID 21355887
- [Result] Gu Z, Li Y, Li H. Use of Condensed Nanofat Combined With Fat Grafts to Treat Atrophic Scars. JAMA Facial Plast Surg. 2018 Mar 1;20(2):128-135. doi: 10.1001/jamafacial.2017.1329. PMID 28975248
- [Derived] Jan SN, Bashir MM, Khan FA, Hidayat Z, Ansari HH, Sohail M, Bajwa AB, Shami HB, Hanif A, Aziz F, Choudhery MS. Unfiltered Nanofat Injections Rejuvenate Postburn Scars of Face. Ann Plast Surg. 2019 Jan;82(1):28-33. doi: 10.1097/SAP.0000000000001631. PMID 30285990